CLINICAL TRIAL: NCT07283393
Title: Observational Prospective Study on Resective and Regenerative Periodontal Therapy: Short & Longterm Follow-up
Acronym: UZFLAPSTUD
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0622
Record Dates: First submitted 2025-11-23; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Periodontal Diseases; Periodontitis
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Periodontitis patients actively treated with regenerative or resective surgery.: Periodontitis patients actively treated with regenerative or resective surgery. The study commences only after the patient has undergone either a regenerative or resective periodontal surgery; the surgical procedure itself is not part of the investigation.
  The objective of the study is to monitor and compare both treatment modalities in the short and long term with respect to tooth survival, bone level, probing pocket depth, tooth sensitivity, mobility, bleeding on probing, and cost-effectiveness.
  The dental patient records will be reviewed to obtain available data from before and during the surgical procedure, including general patient information (age, sex, ASA classification, and medication), periodontal status, radiographic documentation, and clinical photographs.
  Interventions: Diagnostic Test: Periodontal charting, peri-apical radiograph and low-dose small-field cone beam CT

INTERVENTIONS:
Diagnostic Test: Periodontal charting, peri-apical radiograph and low-dose small-field cone beam CT — Clinical measurements through periodontal charting, peri-apical radiography and cone-beam computed tomography. Clinical pictures of the mouth

SUMMARY:
Periodontitis is a common inflammatory disease affecting approximately 40% of the Belgian population.

The goal of this observational study is to learn about the treatment outcomes of surgical periodontal therapy in adults with periodontitis.

The main questions this study aims to answer are:

* Does subsequent surgical intervention further improve periodontal health parameters?
* Is there any significant difference between treatment outcomes of resective and regenerative periodontal surgery.

Participants will:

- Undergo surgical periodontal treatment if residual pocket depth ≥6 mm persists despite good oral hygiene.

Study inclusion was performed after surgical treatment.

- Be screened on various intervals. If there is any recurrent periodontitis, adequate treatment will be performed

In short term, pocket probing depth is our primary outcome and tooth survival is the outcome in the long term.

Secondary outcomes in short-term are bone level, mobility, bleeding on probing, tooth survival and cost-effectiveness.

Long-term outcomes (>5 years) are probing pocket depth, bone level, tooth sensitivity, mobility, bleeding on probing and cost-effectiveness.

DETAILED DESCRIPTION:
Periodontitis is a common condition, affecting approximately 40% of the Belgian populations. The condition most common characteristics are bleeding of the gingiva and bone loss. Left untreated, this disease can lead to severe loss of maxillary or mandibulary bone. Treatment for primary stages of periodontitis don't always require surgical interventions; correction of oral hygiene and deep cleaning the teeth combined, if necessary, with extraction of irrational to treat elements under local anesthesia can be sufficient. Three months after initial treatment, at the re-evaluation, the depth of the tooth pockets, bleeding on probing, mobility and the amount of regression of the gums are reassessed. If the depth of the tooth pockets regressed insuffient, with a depth of at least six milimeters, eventhough the patients oral hygiene is acceptable, further surgical treatment is necessary. A patient is not able to clean these greater pockets.

Resective or regenerative surgery was performed, based on the bone morphology and the patients characteristics.

Inclusion of patients in this study was performed after surgical treatment. Research parameters will be evaluated at 6 months, 1 year, 3 years, 5 years, 7 and 10 years after surgery.

The main questions this study aims to answer are:

* Does subsequent surgical intervention further improve periodontal health parameters?
* Is there any significant difference between treatment outcomes of resective and regenerative periodontal surgery.

Primary outcomes are pocket probing depth in short-term and tooth survival in the long term.

Secondary outcomes in short-term include bone level, mobility, bleeding on probing, tooth survival and cost-effectiveness.

Long-term outcomes (>5 years) are probing pocket depth, bone level, tooth sensitivity, mobility, bleeding on probing and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Min 18 years of age
* Max 6 months since resective or regenerative periodontal surgery
* Good general health

Exclusion Criteria:

* Pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged at least 18 years old have been treated for periodontitis through subgingival debridement. During re-evaluation, remaining pockets were found despite adequate oral hygiene.
  Depending on the anatomy of the defect, resective or regenerative surgery was performed. Patients were included if resective or regenerative periodontal surgery was performed < 6months ago and an informed consent was signed.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Probing depth | At 6 months, 1 year, 3 years, 5 years, 7 years and 10 years of follow-up
  Probing depth evolution in the short term
Tooth retention | From enrollment to the end of the study, at 10 years of follow up
  Survival of tooth in the long-term follow-up

SECONDARY OUTCOMES:
Radiographic bone level | 6 months, 3 years, 5 years, 7 years and 10 years
  A peri-apical radiograph will be taken at various recall appointments. Bone level will be measured using ImageJ software. Calibration will be performed using an orthodontic button, with known dimensions. Two measurements will be made; cemento-enamel junction to the bottom of the pocket and the infra-bony component (alveolar crest to bottom of pocket)
Tooth mobility | At 6 months, 1 year, 3 years, 5, 7 and 10 years of follow-up.
  Mobility of the tooth is assessed using the Miller Classification (1958). Grade 1 is horizontal mobility <1mm, grade 2 is >2mm and grade 3 is horizontal + vertical mobility.
Bleeding on probing | At 6 months, 1 year, 3 years, 5, 7 and 10 years of follow-up
  Bleeding on probing is assessed using a periodontal probe. A probe is inserted in the pocket and bleeding is noted dichotomously.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Long-term follow up of study. No decision yet.